CLINICAL TRIAL: NCT02629705
Title: Investigation of the Effect of Carrageenan as Food Additive on Insulin Resistance in Humans
Brief Title: Study of Carrageenan's Effect on Insulin Resistance in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CGN
Record Dates: First submitted 2015-12-04; First posted 2015-12-14 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Carrageenan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): 1. Placebo intervention
  2. Assessment block (3 days)
  3. Washout-phase of 21-35 days
  4. Carrageenan intervention
  5. Assessment block (3 days)
  Interventions: Dietary Supplement: Carrageenan; Dietary Supplement: Placebo
- Group B (Other): 1. Carrageenan intervention
  2. Assessment block (3 days)
  3. Washout-phase of 21-35 days
  4. Placebo intervention
  5. Assessment block (3 days)
  Interventions: Dietary Supplement: Carrageenan; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carrageenan — Carrageenan 250 mg bid supplemented to a standard food
  Other Names: E407
Dietary Supplement: Placebo — Placebo (Mannitol/Aerosil) bid supplemented to a standard food

SUMMARY:
The purpose of this study is to determine whether the ingestion of the common food additive carrageenan contributes to insulin resistance and thus to the pathogenesis of type 2 diabetes in humans.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) 18.5 - 29.9 kg/m²

Exclusion Criteria:

* any chronic illness
* any ongoing medication
* known infections
* known liver disease
* known renal insufficiency
* alcohol consumption over 30 g/d
* shift work

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-23 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity assessed by oral glucose tolerance test (OGTT): Matsuda index | 2 weeks
Insulin sensitivity assessed by hyperinsulinemic clamp: M-value | 2 weeks

SECONDARY OUTCOMES:
Endogenous glucose production measured by tracer-method | 2 weeks
Cerebral insulin sensitivity measured by MRI | 2 weeks
Intrahepatic triglyceride content | 2 weeks
Glycemia during OGTT | 2 weeks

OTHER OUTCOMES:
Intestinal permeability | 2 weeks
Intestinal microbiome constitution | 2 weeks
Markers of systemic inflammation including lymphocyte activation, cytokines and adipokines | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wagner, M.D, Principal Investigator — University of Tübingen, Department of Internal Medicine
Locations (1):
- University Hospital Tübingen, Department of Internal Medicine, Tübingen, Germany

REFERENCES:
- [Derived] Wagner R, Buettner J, Heni M, Fritsche L, Kullmann S, Wagmuller M, Peter A, Preissl H, Machann J, Jumpertz von Schwartzenberg R, Birkenfeld AL, Pape UF, van Hall G, Plomgaard P, Haring HU, Fritsche A, Thompson KN, Klein R, Stefan N. Carrageenan and insulin resistance in humans: a randomised double-blind cross-over trial. BMC Med. 2024 Nov 26;22(1):558. doi: 10.1186/s12916-024-03771-8. PMID 39593091